CLINICAL TRIAL: NCT04000828
Title: Comparison of Sensimed Triggerfish (TF) 24 Hour Monitoring of the Eye in Glaucoma Patients Before and After Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Katrin Lorenz, Head of clinical trial site, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-14131
Record Dates: First submitted 2019-05-27; First posted 2019-06-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single Arm (Other): all patients receive the measurement with Sensimed Triggerfish
  Interventions: Device: Placement of Sensimed Triggerfish

INTERVENTIONS:
Device: Placement of Sensimed Triggerfish — Sensimed Triggerfish is placed on the corneal surface

SUMMARY:
A 24 hour profile is recorded using Sensimed Triggerfish in glaucoma patients before and after Trabecuelctomy

ELIGIBILITY:
Inclusion Criteria:

* Patient must have the willingness and ability to provide signed informed consent
* Patient is able to comply with the study procedure
* Patient must be ≥ 18 years old
* Diagnosis of primary open angle glaucoma (EGS criteria) including pseudoexfoliation glaucoma/ normal tension glaucoma/ pigmentary glaucoma in the study eye
* planned trabeculectomy in the study eye
* in preparation for trabeculectomy, all preoperative IOP lowering medication has been replaced by Dorzolamid 20 mg/ml + Timolol 5mg/ml preservative free eye drops in the study eye for at least 28 days before Triggerfish® profile
* Patient has consented to be in the trial and signed informed consent is available before any study related procedures are carried out
* Visual Acuity of 20/200 or better in both eyes
* Ability of subject to understand the character and individual consequences of the study

Exclusion Criteria:

* Subjects with contraindications for wearing contact lenses in the study eye
* secondary glaucoma in the study eye
* History of refractive surgery in the study eye
* History of intraocular surgery in the last three months in the study eye
* Severe dry eye syndrome as judged by the investigator in the study eye
* Keratoconus or other corneal abnormalities
* Any other abnormality in the study eye, that prevents the safe placement of the device after investigators decision
* Conjunctival or intraocular inflammation in the study eye
* Simultaneous participation in other clinical trials
* Previous IOP-lowering intervention in the study eye
* Current shift workers (applicable for at least 3 months)
* Transmeridian flight < 2 months before screening (6 hours time shift)
* Subjects with pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Amplitude | up to 14 weeks
  Comparison of Amplitude between the preoperative Triggerfish Profile and the Triggerfish Profile three months after Trabeculectomy

SECONDARY OUTCOMES:
Correlation of other parameters | up to 14 weeks
  Correlation of IOP and Triggerfish Profile, Correlation of IOP, blood pressure and heart rate, Evaluation of 24 hours nyctohemeral rhythm of measurements before and after trabeculectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Department of Ophthalmology, University Medical Center Johannes Gutenberg University Mainz, Mainz, Germany